CLINICAL TRIAL: NCT02345681
Title: Impact of Rational Control of Fluid Balance in the Intensive Care Unit.IRIHS-REA
Brief Title: Impact of Rational Control of Fluid Balance in the Intensive Care Unit
Acronym: IRIHS-REA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC14_0268
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Fluid Balance of ICU Patients; Fluid Overload
Keywords: furosemide; under strict conditions; normalize; ICU patients; fluid balance
MeSH Terms: conditions — Edema | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Test Furosemide (Experimental): We will test our furosemide algorithm in one arm
  Interventions: Drug: Furosemide
- Classical Strategy (No Intervention): It's a classical strategy without diuretics

INTERVENTIONS:
Drug: Furosemide
  Arms: Test Furosemide

SUMMARY:
Patients admitted in the Intensive Care Unit (ICU) frequently display and excessive fluid balance over a very short period of time. This positive fluid balance is the consequence of different organ failures (pulmonary, cardio-vascular, kidney…) or aggressive fluid resuscitation, which is mandatory in the early phase of ICU course. However recent data strongly suggest that an excessive fluid balance could be detrimental per se (increase of ICU morbidity or even mortality). There are controversies regarding the potential benefit of controlling this fluid balance with diuretics which are commonly used worldwide in various indications (acute and chronic heart failure, chronic kidney failure). In the ICU literature data are lacking, regarding the possible advantages and drawbacks of diuretics in this indication. The aim of our study is to test an algorithm with furosemide to reduce fluid overload in severe ICU-patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or more
* Patients receiving endo-tracheal intubation and mechanical ventilation during their stay in the ICU
* Weight increase of at least 3 % during the stay. Baseline weight is regarded as the weight at the 24th hour after ICU admission
* FiO2 < 60 %, PEEP < 10cmH20
* No administration of catecholamines other than dobutamine at a dose of 10 microg.Kg-1.min-1

Exclusion Criteria:

* Pregnancy
* Patient with a moribund state at ICU arrival
* Acute brain injury (traumatic brain injury, subarachnoid hemorrhage, intra-cerebral bleeding, stroke, meningo-encephalitis, coma from medication origin)
* Chronic kidney disease defined as creatinin clearance < 30mL.min-1 and/or with chronic dialysis
* Mandatory administration of diuretics (cardiogenic pulmonary oedema, LVEF < 30 %)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Evolution of fluid balance between randomisation and extubation (fluid balance in our study = Patient's weight at randomisation - Patient's initial weight (Kg) defined as the weight at admission) | Day 60
  Definition of fluid balance in our study = Patient's weight at randomisation - Patient's initial weight (Kg) defined as the weight at admission

SECONDARY OUTCOMES:
Number of ventilatory-free days | Day 28
Number of ICU-free days | Day 60
Period of mechanical Ventilation | Day 60
Extubation Failure | Day 60
ICU Period of stay | Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Karim Asehnoune, Principal Investigator — Nantes University Hospital; Christine LEBERT, Principal Investigator — CHD La Roche sur Yon
Locations (3):
- France (3):
  - Hôpital François Mitterand, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - CHU de Nantes, Nantes

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152
- [Derived] Cinotti R, Lascarrou JB, Azais MA, Colin G, Quenot JP, Mahe PJ, Roquilly A, Gaultier A, Asehnoune K, Reignier J. Diuretics decrease fluid balance in patients on invasive mechanical ventilation: the randomized-controlled single blind, IRIHS study. Crit Care. 2021 Mar 10;25(1):98. doi: 10.1186/s13054-021-03509-5. PMID 33691730